CLINICAL TRIAL: NCT04343443
Title: Acute Heart Failure With Reduced Ejection Fraction - COngestion Discharge Evaluation: Evaluation de la Congestion à la Sortie d'Hospitalisation Pour Insuffisance Cardiaque aiguë à Fraction d'éjection altérée ou modérément altérée
Brief Title: Acute Heart Failure With Reduced Ejection Fraction - COngestion Discharge Evaluation
Acronym: AHF-CODE-R
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pr. Nicolas GIRERD, Acute Heart Failure With Reduced Ejection Fraction - COngestion Discharge Evaluation: Evaluation de la Congestion à la Sortie d'Hospitalisation Pour Insuffisance Cardiaque aiguë à Fraction d'éjection altérée ou modérément altérée, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019PI188-3
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-03

CONDITIONS: Acute Heart Failure
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients hospitalized for acute heart failure (Other): Patients hospitalized for acute heart failure will undergo the following evaluations:
  * Clinical examination centered on congestion
  * Cardiopulmonary , peritoneal , jugular and renal venous Doppler ultrasounds
  * Blood sample retrieved for biological assessment and biobanking
  * Telephone interview
  Interventions: Procedure: Clinical examination centered on congestion; Procedure: Cardio-pulmonary, peritoneal, jugular and renal Doppler ultrasounds and liver elastography; Procedure: Biological: Blood sample retrieved for biological assessment and biobanking; Procedure: Telephone interview; Behavioral: Kansas City Cardiomyopathy Questionnaire (KCCQ)

INTERVENTIONS:
Procedure: Clinical examination centered on congestion — Clinical examination centered on congestion (ASCEND, NYHA and Ambrosy Score) will be performed before discharge from hospital
Procedure: Cardio-pulmonary, peritoneal, jugular and renal Doppler ultrasounds and liver elastography — Cardio-pulmonary, peritoneal, jugular and renal Doppler ultrasounds and liver elastography will be performed before discharge from hospital
Procedure: Biological: Blood sample retrieved for biological assessment and biobanking — Blood sample collection will be performed before discharge from hospital
Procedure: Telephone interview — Telephone interview will be performed at 3, 12 months and 24 months after discharge from hospital
Behavioral: Kansas City Cardiomyopathy Questionnaire (KCCQ) — Questionnaire centered on patient's quality of life at discharge and 3, 12 and 24 months after discharge

SUMMARY:
The AHF-CODE reduced study is a prospective, non-randomized, monocenter study performed in patients with heart failure with reduced ejection fraction admitted for worsening heart failure.

The main objective of the AHF-CODE study is to identify congestion markers (clinical, biological and ultrasound) at the end of hospitalization for acute heart failure that are associated with the risk of all cause death or rehospitalization for acute heart failure within 3 months of hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalised for acute heart failure.
* Patients with reduced ejection fraction (Ejection Fraction <40%) or (40% ≤ Ejection Fraction < 50)
* Patients considered clinically discharging from hospitalisation for acute heart failure.
* Age ≥18 years
* Patients having received complete information regarding the study design and having signed their informed consent form.
* Patient affiliated to or beneficiary of a social security scheme.

Exclusion Criteria:

* Comorbidity for which the life expectancy is ≤ 3 months
* Dialysis patient (peritoneal dialysis or hemodialysis) or patients with glomerular filtration rate <15 ml/min/m2 at inclusion.
* History of lobectomy or pneumonectomy lung surgery
* Severe pulmonary or pleural pathology preventing reliable acquisition of lung ultrasound images: severe emphysema, chronic pleurisy, pulmonary fibrosis, etc.
* Pregnant woman, parturient or nursing mother
* Adult person subject to a legal protection measure (guardianship, curatorship, safeguard of justice) Adult person who is unable to give consent
* Person deprived of liberty by a judicial or administrative decision,
* Person subject to psychiatric care pursuant to Articles L. 3212-1 and L. 3213-1 of the Public Health Code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-08-21 (Actual); Primary Completion 2026-08-21 (Estimated); Study Completion 2028-08-21 (Estimated)

PRIMARY OUTCOMES:
Rate of all-cause death | 3 months after hospital discharge
  composite endpoint: rate of all-cause death, hospitalization for acute heart failure or day-hospital IV diuretics injection for acute HF during 3 months following day hospitalization (with outcome 2 and 3)
Rate of re-hospitalisation for acute heart failure | 3 months after hospital discharge
  composite endpoint: rate of all-cause death, hospitalization for acute heart failure or day-hospital IV diuretics injection for acute HF during 3 months following day hospitalization (with outcome 1 and 3)
Rate of day-hospital or in-home IV diuretics injection for acute HF | 3 months after hospital discharge
  composite endpoint: rate of all-cause death, hospitalization for acute heart failure or day-hospital IV diuretics injection for acute HF during 3 months following day hospitalization (with outcome 1 and 2)

SECONDARY OUTCOMES:
Rate of all-cause death | 3, 12 and 24 months after hospital discharge
Rate of re-hospitalisation for acute heart failure | 3, 12 and 24 months after hospital discharge
Rate of day-hospital IV diuretics injection for acute HF | 3, 12 and 24 months after hospital discharge
Rate of all-cause death | 3, 12 and 24 months after hospital discharge
  composite endpoint : Rate of all-cause death or hospitalisation for acute heart failure at 3, 12 and 24 months after hospital discharge (with outcome 8)
Rate of hospitalisation for acute heart failure | 3, 12 and 24 months after hospital discharge
  composite endpoint : Rate of all-cause death or hospitalisation for acute heart failure at 3, 12 and 24 months after hospital discharge (with outcome 7)
Rate of all-cause death | 3, 12 and 24 months after hospital discharge
  composite endpoint: Rate of all-cause death or hospitalisation for acute heart failure at 3, 12 and 24 months after hospital discharge (with outcome 10)
Rate of hospitalisation for acute heart failure | 3, 12 and 24 months after hospital discharge
  composite endpoint: Rate of all-cause death or hospitalisation for acute heart failure at 3, 12 and 24 months after hospital discharge (with outcome 9)
NYHA (New York Heart Association) class | 3, 12 and 24 months after hospital discharge
Natriuretic peptides | At inclusion
  BNP or Nt-Pro BNP
Renal function assessed by glomerular filtration rate | At inclusion
Plasma volume | At inclusion
  calculated from haemoglobin and haematocrit value
Blood potassium | At inclusion
Rate of all-cause death | 3, 12 and 24 months after hospital discharge
  composite endpoint: Rate of all-cause death or hospitalisation for acute heart failure at 3, 12 and 24 months after hospital discharge (with outcome 17)
Rate of hospitalisation for acute heart failure | 3, 12 and 24 months after hospital discharge
  composite endpoint : Rate of all-cause death or hospitalisation for acute heart failure at 3, 12 and 24 months after hospital discharge (with outcome 16)
Liver elastography value | At inclusion
  Measured with Fibroscan®
Quality of life assessed by Kansas City Cardiomyopathy Questionnaire | At inclusion and 3, 6 and 24 months
  Assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Vandœuvre-lès-Nancy, France